CLINICAL TRIAL: NCT01429168
Title: The Randomized Etoricoxib Study in Patients With Osteoarthritis Not Responding to Analgesic Drugs - THE RESPOND-EUROPE STUDY
Brief Title: A Study of Etoricoxib in Participants With Osteoarthritis Not Responding to Analgesic Drugs (MK-0663-142)
Acronym: RESPOND-EUROPE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-142
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: All Enrolled Participants (Experimental): All participants will receive open-label etoricoxib 60 mg orally daily during Part 1.
  Interventions: Drug: Etoricoxib
- Part 2: Etoricoxib (Experimental)
  Interventions: Drug: Etoricoxib
- Part 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo for etoricoxib

INTERVENTIONS:
Drug: Etoricoxib — One 60-mg tablet orally daily
  Other Names: MK-0663
  Arms: Part 1: All Enrolled Participants; Part 2: Etoricoxib
Drug: Placebo for etoricoxib — One 60-mg tablet orally daily
  Arms: Part 2: Placebo

SUMMARY:
This two-part study will evaluate the effectiveness of etoricoxib in controlling pain in participants with osteoarthritis who are experiencing inadequate response to their current treatments. In Part 1, all participants will receive open-label etoricoxib 60 mg daily. Those participants who experience a clinically meaningful response to etoricoxib 60 mg daily within two weeks will be eligible to enter the double-blind withdrawal period (Part II). Responders entering Part 2 will be randomized in a 1:1 ratio to receive either etoricoxib 60 mg or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis of the knee or hip that requires treatment
* American Rheumatism Association (ARA) functional Class I, II or III
* Receiving a stable dose of a traditional non-steroidal anti-inflammatory drug (NSAID), a Cox-2 selective inhibitor (other than etoricoxib, e.g. celecoxib), opioid therapy or tramadol to treat their osteoarthritis-related pain for at least 2 weeks and willing to maintain treatment during baseline phase
* Moderate to severe daily pain intensity on his or her current pain regimen
* Excepting osteoarthritis, patient is judged to be in otherwise general good health based on medical history, physical examination, and routine laboratory tests
* Negative serum pregnancy test

Exclusion Criteria:

* Has not experienced at least 3 consecutive days of daily pain intensity >4 on 10-point scale
* Severe hepatic insufficiency
* Advanced renal insufficiency
* Presence of gastro-intestinal ulcer disease with active bleeding or history of the same within the past 6 months or a presence or history of inflammatory bowel disease
* History of gastric, biliary (including gastric bypass surgery), or small intestinal surgery that results in clinical malabsorption
* Receiving or will likely require treatment with ≥14 consecutive days or repeated courses of pharmacologic doses of corticosteroids
* Established ischemic heart disease, peripheral arterial disease, and/or cerebrovascular disease including a history of stroke, myocardial infarction or transient ischemic attack, and recent revascularization procedures
* Any other contraindications mentioned in the approved study drug European Union (EU) Summary of Product Characteristics (SmPC)
* Therapy with glucosamine and/or chondroitin sulfate for <6 months prior to study start.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Mean Time to Loss of Efficacy in the Double Blind Withdrawal Period (Part 2) | Week 3 to Week 7

SECONDARY OUTCOMES:
Proportion of Participants who Achieve ≥30% Reduction in Pain During Part I | Week 1 to Week 3
Change in Mean of Daily Pain Scores | Week 1 to Week 7
Proportion of Participants Meeting Criteria for Loss of Efficacy in Part 2 | Week 3 to Week 7